CLINICAL TRIAL: NCT05921786
Title: Record Voxel Rate Nonlinear Optical Microscope to Unravel Brain Connectome and Signaling-Establish Reliably Electrophysiological Readouts From Human-induced Pluripotent Stem Cells (hiPSCs)-Derived Cerebral Organoids and Surgically Dissected Human Live Brains
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202302097RIND
Record Dates: First submitted 2023-06-18; First posted 2023-06-27 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-05

CONDITIONS: Brain Diseases; Brain Tumor
Keywords: brain diseases, brain tumor
MeSH Terms: conditions — Brain Diseases; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiphoton microscopy (Experimental)
  Interventions: Device: Multiphoton microscope
- Electrophysiological system (Experimental)
  Interventions: Device: Electrophysiological system

INTERVENTIONS:
Device: Electrophysiological system — Electrophysiological system is used for examining voltage variation in biological samples. And multiphoton microscopy is a common type of nonlinear optical microscope.
  Arms: Electrophysiological system
Device: Multiphoton microscope — Multiphoton microscope acquires high-resolution image based on nonlinear optics and can be used for detect biological specimens.
  Arms: Multiphoton microscopy

SUMMARY:
The research aims to establish a big database of multiple kinds of brain tissues and prove the relevance of human brain tissue models and hiPSCs-derived organoid models.

DETAILED DESCRIPTION:
Brain diseases are very difficult diseases to treat, and when developing related medical cures for saving lives, however, it is difficult to obtain examining samples, especially like normal brain tissue since it is necessary to preserve the brain tissue of patients to ensure its functionality. Among the numerous brain diseases, there are many diseases that combine surgery, chemotherapy, and immunotherapy in treatment. For example, for brain tumors, surgery is the most important treatment that can effectively prolong the survival time of patients. Numerous neurological functions, tumors generated in such important organs, require careful judgment of resection strategy in surgical treatment. In addition to achieving complete tumor resection, subsequent chemotherapy and immunotherapy are also important factors to improve prognosis. Traditionally, the neurosurgeon's experience and various preoperative examinations are used to judge the type and distribution of the disease, which may lead to inconsistent results due to different personal experiences. The current methods that can be used clinically to help improve the integrity of resection (such as intraoperative fluorochrome and intraoperative magnetic resonance imaging) are relatively indirect methods of judgment, but it is hard to directly know the detailed information of the disease before surgery, and the assessment results of formalin-fixed paraffin-embedded (FFPE) section through the standard operation of pathological procedures are used to formulate drug treatment strategies, which may greatly affect the prognosis of patients. According to the current intraoperative cryopathology, there are many brain tumors that cannot be classified easily by it. When searching the literature, there are also few related studies that try to solve this problem, but in addition to the insufficient sample size, it is also impossible to acquire appropriate conclusions due to the limited number of samples. Therefore, through this study, we want to implement optical microscopy and electrophysiological analysis system to capture images and electrophysiological signals of some remaining brain diseased tissues after surgical resection, and compare the acquired datas with the results obtained from human brain organoid tissues. Eventually, construct a large database of brain tissue can also verify whether human brain organoids can completely compare with real human brain samples can truly improve the medical operation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than the age of 18 with diagnosis of brain disease (both newly-diagnosed or recurrent) who are suitable and willing to receive resection surgery.

Exclusion Criteria:

1. Patients who cannot give consent to participate in the study.
2. The tumor samples failed to give a conclusive pathological diagnosis by standard pathological workflow.
3. Patients who only receives biopsy surgery rather than resection surgery.
4. Significant post-irradiation effect or radiation necrosis reported in the pathological examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Acquire neuronal structual (image frame) results of different brain regions | 3 years
  By interpreting the microscopic images of different brain regions' tissues , an attempt is made to understand the structure of brain disease tissues (via cell morphology, microvessels, etc).
Acquire electrophysiological readout (voltage amplitude, mV) datas of different brain regions | 3 years
  By interpreting the neuron electric reactive datas, an attempt is made to know the neuronal activity (via detecting voltage amplitude change) between multiple neurons.

SECONDARY OUTCOMES:
To conduct imaging for multiple types of human brain tissues and construct the neuron image database | 3 years
  Accumulating the microscopic images and neuron electrosiological signals, the image database of normal and diseased neuron reaction can be constructed.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, National Taiwan University Hospital and College of Medicine, National Taiwan University, Taipei, Taiwan